CLINICAL TRIAL: NCT04394260
Title: Equality in Caregiving: Facilitating Caregiver Mastery Among LGBT Caregivers of PLWD
Acronym: EIC
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Whitney Wharton, Associate Professor, Emory University
Other Study IDs: STUDY00002246; IRB00113264 (Other: Emory University); 5P30AG064200-02 (NIH)
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Dementia; Caregiver Burnout
Keywords: Person Living with Dementia (PLWD); Lesbian, Gay, Bisexual, Transgender (LGBT); Informal caregiver; Savvy Caregiving Program; Alzheimer's Disease (AD); Alzheimer's Disease and Related Dementias (ADRD)
MeSH Terms: conditions — Dementia; Caregiver Burden; Homosexuality, Female; Homosexuality; Bisexuality; Alzheimer Disease | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LGBT Caregivers Participating in a Focus Group: LGBT caregivers attending a focus group after watching the videos of the remote learning Savvy Caregiver Program. The focus group will guide modification of the Savvy Caregiver Program to meet the needs of LGBT caregivers of PLWD.
  Interventions: Behavioral: Savvy Caregiver Program via Remote Learning; Behavioral: Focus group

INTERVENTIONS:
Behavioral: Savvy Caregiver Program via Remote Learning — The SCP program is comprised of four pre-recorded Savvy Caregiver videos (each 1 hour and 45 minutes in length). Course material was designed to provide informal caregivers with the knowledge, skills, and attitude needed to carry out their role as a caregiver for a person living with dementia (PLWD). Course learning objectives include: 1) introduction to dementing disorder; 2) caregiver self-care; 3) the anchors of enjoyable involvement; 4) levels of thinking and performance; 5) strengthening the family as a resource for caregiving; and 6) review and integration of the previous sections.
  Other Names: Savvy Caregiver Program provided via Pre-Recorded Video
Behavioral: Focus group — After watching the Savvy Caregiver videos participants will take part in a focus group to discuss their experience with the SCP and how the course material applies to them as a LGBT caregiver. The semi-structured discussion will include, but not be limited to the following questions: 1) Can you tell me about your role as a caregiver? (Probes: living situation, experiences, challenges). 2) What went well with the SCP, and what could be improved? 3) How relevant to your situation as an LGBT caregiver were the course materials? 4) How well did the questionnaire reflect your experiences with discrimination due to sexual orientation and/or gender identity? (Probe about when working with your care recipient's health care providers, in-home aides/visiting nurses, adult day care staff, respite, etc? 5) What are some of the additional caregiver challenges that should be considered in these questionnaires? (Probes: mental health, physical health, and social life strain, Quality of life, stress).

SUMMARY:
The goal of this study is to adapt existing Savvy Caregiving Program (SCP) for lesbian, gay, bisexual, transgender (LGBT) caregivers of person living with dementia (PLWD). After watching the SCP Remote Learning videos, participants will attend a focus group to discuss how the program could be changed to meet the specific needs of LGBT caregivers of PLWD.

DETAILED DESCRIPTION:
Over 15 million family caregivers provide more than $200 billion in unpaid care to a person living with dementia (PLWD). This dynamic has been shown to influence the PLWD, as well as the physiological and psychological health of the caregiver. Depression and stress have been linked to caregiving, and both are independent risk factors for dementia. In addition to subjective indices of stress and depression, stress biomarkers have been shown to be higher in dementia caregivers vs. non-caregivers.

The complex caregiving experience depends on many factors, including the disease state of the PLWD, the nature of the relationship (spouse vs. child vs. friend), as well as the race, ethnicity, gender identity, and sexual orientation of the individuals involved. Informal caregiving for PLWD by lesbian, gay, bisexual, and transgender (LGBT) individuals continues to receive limited attention, and current research rarely examines how caregiving for PLWD affects the LGBT community. Estimates of the number of LGBT adult caregivers range from 27% to more than 45%.

Although the National Institutes of Health and the Institute of Medicine have recently emphasized the disparity in LGBT aging issues, little is known about stress experienced by LGBT caregivers compared with non-LGBT caregivers. Research with LGBT caregivers of PLWD has shown that they experience higher rates of physical, emotional, and financial strain, and are more likely to help with medical/nursing tasks. Higher levels of LGBT caregiver stress may be due to the fact that LGBT caregivers are less likely to seek out supportive services or disclose their LGBT identities. Higher rates of caregiving stress for LGBT caregivers may stem from years of stigma and failure of current interventions and resources to assess the unique stressors of LGBT persons adequately. Fear of discrimination, denial of services, and receiving poor-quality services may also contribute to reluctance to seek assistance. Moreover, LGBT persons are more likely to suffer from behavioral, psychological and physiological health issues than non-LGBT persons, all of which are independent predictors of Alzheimer's disease and related dementias (ADRD).

The Savvy Caregiver Program (SCP) was developed by Kenneth Hepburn PhD to train informal caregivers of community dwelling PLWD. The SCP consists of educational instruction and in-class exercises that engage participants on a functional level. Course material was designed to provide informal caregivers with the knowledge, skills, and attitude needed to carry out their role as a caregiver for a PLWD. The existing SCP is comprised of weekly, two-hour interactive classes, over six consecutive weeks. Dr. Hepburn and his team also created four, one hour and 45 minute long, videos to be used as a method of remote learning that cover the same material as the in-person program. These videos will be used in this study.

The primary goal of this study is to adapt the SCP to address the context-specific challenges faced by LGBT informal caregivers of PLWD, in preparation for a larger efficacy trial. The researchers will conduct focus groups to engage LGBT caregivers and a LGBT Community Advisory Board in the process of adapting the existing SCP to their needs.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as an LGBT adult (18 yrs and over)
* Providing informal care to a community dwelling adult family member or friend for at least 3 months OR
* Was formerly providing informal care to a community dwelling adult family member or friend for at least 6 months no more than 5 years ago
* Willing to participate in a one hour survey
* Agree to participate in up to 12 hours of clinical trial activities, including up to 6 hours of videos

Exclusion Criteria:

• Any significant diagnosed systemic illness or unstable diagnosed medical condition that could affect cognition (i.e. MCI), cause difficulty complying with the protocol or consenting for study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identification as a LGBT adult
Study Population: Lesbian, gay, bisexual, transgender (LGBT) caregivers of person living with dementia (PLWD)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Development of SCP for LGBT Caregivers of PLWD | Day of Focus Group (Day 1)
  A version of the SCP will be developed to meet the needs of LGBT Caregivers of PLWD through focus groups discussing the SCP after participants watch all of the videos. Semi-structured discussions in the focus group will include, but not be limited to the following questions: 1) Can you tell me about your role as a caregiver? 2) What did you like about the SCP, and what could be improved? 3) How relevant to your situation as an LGBT caregiver were the course materials? 4) How well did the questionnaire reflect your experiences with discrimination due to sexual orientation and/or gender identity? 5) What are some of the additional caregiver challenges that should be considered in these questionnaires?

CONTACTS AND LOCATIONS:
Overall Officials: Whitney Wharton, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Goizueta Alzheimer's Disease Research Center (ADRC), Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlies the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared
Supporting Information: ICF
Time Frame: Immediately following publication with no end date
Access Criteria: Researchers who provide a methodologically sound proposal to achieve aims in the approved proposal will get access. Proposals should be directed to (w.wharton@emory.edu). To gain access, data requestors will need to sign a data access agreement. Data will then be shared directly via csv or excel file.